CLINICAL TRIAL: NCT03624088
Title: Understanding Social, Cultural, and Religious Factors Influencing BRCA Genetic Testing in the Orthodox Jewish Community
Brief Title: CBPR - BRCA Genetic Testing Among Orthodox Jews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Katherine D. Crew, Associate Professor of Medicine and Epidemiology at the Columbia University Medical Center, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAO1760
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Prevention; Genetic Testing; Orthodox Jewish; Community-Based Participatory Research; BRCA; Decision Support
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Intervention (Experimental): Participants will complete a baseline questionnaire. They will then self-administer the web-based decision aid, RealRisks. Upon completion, they will complete two more surveys: one within 1 month of completing RealRisks and one six months after completing RealRisks.
  Interventions: Behavioral: RealRisks

INTERVENTIONS:
Behavioral: RealRisks — RealRisks is a web-based patient decision aid with modules on risk assessment, family history and breast cancer, genetic testing, and prevention options. Participants enter family history data into RealRisks, and RealRisks calculates 5-year breast cancer risk, lifetime breast cancer risk, and the probability of carrying a BRCA mutation. This information is then interactively presented to the participant. RealRisks facilitates the participant in identifying their intention to undergo BRCA genetic testing and the factors that are important to the participant in making this decision. RealRisks produces a summary of all of this information that the participant can print and take with her to a health care appointment.
  Other Names: RealRisks Decision Aid

SUMMARY:
This study evaluates a web-based decision aid, named RealRisks, in promoting genetic testing intention among Orthodox Jewish women. 50 Orthodox Jewish women will take a baseline survey, self-administer the decision aid, and then complete two more surveys: one within one month of completing the decision aid and one at 6 months after completing the decision aid.

DETAILED DESCRIPTION:
Breast cancer confers significant morbidity and mortality on women in the U.S. and ovarian cancer is the most lethal gynecologic malignancy. Genetic determinants, such as germline mutations in the BRCA1 and BRCA2 genes, confer the greatest impact on breast and ovarian cancer risk. Hereditary breast and ovarian cancer syndrome (HBOC) is an inherited condition that is most commonly associated with mutations in the BRCA1 and BRCA2 genes. An estimated 2-7% of breast cancers and 10-15% of ovarian cancers result from inherited mutations in BRCA1 and BRCA2. Mutation carriers have lifetime risks of breast and ovarian cancer of 40-60% and 20-40%, respectively.

The prevalence of three founder mutations in the BRCA1 and BRCA2 genes is up to 2.5% among Ashkenazi Jews and genetic testing for this 'founder' panel is relatively inexpensive. About 1 in 40 individuals of Ashkenazi (central and eastern European) Jewish descent carry a founder mutation in the BRCA1 (5382insC or 185delAG) or BRCA2 (6174delT) genes. Based upon U.S. PreventiveServices Task Force guidelines, Ashkenazi Jewish women with any first- or second-degree relatives with breast or ovarian cancer should be referred for BRCA genetic counseling.

The perceived benefits and risks of genetic testing may vary by demographic, cultural, and religious backgrounds. Orthodox Jews often consult with Rabbinic and communal authorities in medical decision-making, which is consistent with their religious values. The Jewish community is already familiar with genetic testing due to successful testing programs for genetic disorders, such as Tay-Sachs, an autosomal recessive disease. However, there are unique challenges to testing for BRCA genes, which are inherited in an autosomal dominant fashion and predispose to adult-onset diseases, such as breast and ovarian cancer.

This study will test the efficacy of a patient-centered, web-based decision aid called RealRisks in a pilot study of 50 Orthodox Jewish women, using a pre-/post-test design. Genetic testing intention will be assessed at baseline, within 1 month after exposure to RealRisks, and at 6 months. This pilot study will allow the investigator to determine an effect size that can be used to design a well-powered randomized controlled trial in the future.

The ultimate goal is to understand social, cultural, and religious factors influencing BRCA genetic testing in the Orthodox Jewish community.

ELIGIBILITY:
Inclusion Criteria:

* >= 25 years of age
* Completed a previous cross-sectional survey and agreed to future contact
* Eligible for BRCA testing based on Six Point Scale

Exclusion Criteria:

* Personal history of breast or ovarian cancer
* Prior genetic counseling or genetic testing for BRCA mutations
* Participated in previous RealRisks workshop

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 50 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Change in proportion of participants who intend to undergo or have completed genetic testing compared to baseline | 1 month
  Question assessing subject's intention of undergoing genetic testing or completion of genetic testing

SECONDARY OUTCOMES:
Change in proportion of participants who make an informed choice about getting BRCA genetic testing. | 1 month, 6 months
  The degree to which a decision is based on relevant, good quality information, and reflects the decision-maker's values. Calculated using knowledge and attitude scores: to be an informed choice, a patient needs a sufficient knowledge score and a decision that is consistent with their attitude score

OTHER OUTCOMES:
Change in proportion of participants who have accurate breast cancer risk perception | 1 month, 6 months
  5 questions assessing subject's perceived risk of developing breast cancer on a relative and numeric scale
Change in proportion of participants who describe experiencing significant breast cancer worry | 1 month, 6 months
  2 questions on a 7-point Likert scale assessing breast cancer worry
Change in BRCA testing knowledge | 1 month, 6 months
  11 true/false questions to assess knowledge about HBOC genetic testing
Change in proportion of participants who report positive attitudes towards BRCA genetic testing | 1 month, 6 months
  4 items to assess attitudes towards genetic testing
Proportion of patients who experience decision conflict | Baseline, 1 month, 6 months
  10 question scale to assess decision conflict regarding genetic testing
Proportion of patients who experience decisional regret | 6 months
  5 items rated on a 5-point Likert scale to assess views about genetic testing decision
Change in decision autonomy regarding BRCA testing | 1 month
  15 questions rated on a 7-point Likert scale to assess autonomous self-regulation of health-related behaviors
Change in decision self-efficacy regarding BRCA testing | 1 month
  11 questions rated on a 5-point Likert scale to assess decision self-efficacy on genetic testing
Change in Perceived BRCA mutation risk | 1 month, 6 months
  5-point Likert scale assessing patient's perceived risk of carrying HBOC mutation
Perception of stigma associated with carrying BRCA mutation | Baseline, 1 month, 6 months
  8 questions rated on a 7-point Likert scale assessing stigma related BRCA genetic testing

CONTACTS AND LOCATIONS:
Overall Officials: Katherine D Crew, MD, MS, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trivedi MS, Manley H, Yi H, Silverman T, Chung WK, Appelbaum PS, Starck R, Schecter I, Kukafka R, Crew KD. Pilot study of a decision aid on BRCA1/2 genetic testing among Orthodox Jewish women. Fam Cancer. 2024 Nov;23(4):491-498. doi: 10.1007/s10689-024-00371-6. Epub 2024 Apr 12. PMID 38609522